CLINICAL TRIAL: NCT03252249
Title: Duration of Dual Anti-Platelet Therapy in Acute Coronary Syndrome
Brief Title: Duration of Dual Anti-Platelet Therapy (DUAL-ACS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC16104
Record Dates: First submitted 2017-08-09; First posted 2017-08-17 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2023-11

CONDITIONS: Acute Coronary Syndrome; Coronary Artery Disease
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease | interventions — Dual Anti-Platelet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 months dual anti-platelet therapy (Active Comparator): 3 months dual anti-platelet therapy.
  Interventions: Other: 3 months dual anti-platelet therapy
- 12 months dual anti-platelet therapy (Active Comparator): 12 months dual anti-platelet therapy.
  Interventions: Other: 12 months dual anti-platelet therapy

INTERVENTIONS:
Other: 3 months dual anti-platelet therapy — Patients with acute coronary syndrome will be randomised to 3 months dual anti-platelet therapy.
  Arms: 3 months dual anti-platelet therapy
Other: 12 months dual anti-platelet therapy — Patients with acute coronary syndrome will be randomised to 12 months dual anti-platelet therapy.
  Arms: 12 months dual anti-platelet therapy

SUMMARY:
Despite substantial evidence supporting the use of dual anti-platelet therapy in patients with acute coronary syndrome, there remains major uncertainty regarding the optimal duration of therapy. Recent evidence suggests that shorter durations of dual anti-platelet therapy are superior because the avoidance of atherothrombotic events is counterbalanced by the greater risks of excess major bleeding with apparent increases in all-cause mortality with longer durations. We here propose an international randomised controlled trial of 18,318 patients with type 1 myocardial infarction allocated to differing durations of dual anti-platelet therapy. We will use electronic health record linkage to track duration of therapy and clinical outcomes in a real-world, real-time, efficient and highly cost-effective trial. This has the potential to define treatment duration, settle a major outstanding international controversy, and influence modern cardiology practice across the world.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Clinical diagnosis of Type 1 myocardial infarction within 12 weeks
* In the opinion of the attending clinician requires dual anti-platelet therapy with aspirin and a P2Y12 receptor antagonist
* Resident in the country of recruitment with their unique health identifier
* The attending clinician has equipoise regarding the duration of therapy
* Provision of informed consent

Exclusion Criteria:

* Clear indication for specific duration of dual anti-platelet therapy
* Type 2 myocardial infarction
* Contraindication to aspirin or P2Y12 receptor antagonist
* Non-resident in the country of recruitment
* Previous recruitment into the trial
* Inability or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5094 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2023-02-04 (Actual); Study Completion 2023-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Newby, Principal Investigator — University of Edinburgh
Locations (1):
- Edinburgh Royal Infirmary, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All randomised participants in database.
Pre-assignment Details: 42 participants were excluded from the ITT population following randomisation, those who subsequently became ineligible after a diagnosis other than Type 1 myocardial infarction (MI) and withdrawn from the trial were excluded.
Period: Overall Study
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Started | 2526 | 2526
Completed | 2526 | 2526
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy | Total
Number analyzed (Participants) | 2526 | 2526 | 5052
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing data
  years
    number analyzed (Participants) | 2522 | 2522 | 5044
    (all) | 63.4 (10.9) | 63.4 (10.8) | 63.4 (10.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex; Female, Male: Female | 684 | 685 | 1369
  Sex; Female, Male: Male | 1838 | 1837 | 3675
  Sex; Female, Male: Not available | 4 | 4 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 285 | 284 | 569
  Mixed | 1 | 2 | 3
  Asian | 12 | 18 | 30
  Black | 2 | 1 | 3
  Other | 7 | 2 | 9
  Not stated or not known | 50 | 54 | 104
  Missing | 5 | 1 | 6
  Data not collected for Scotland or New Zealand | 2164 | 2164 | 4328
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2265 | 2269 | 4534
  New Zealand | 261 | 257 | 518
Social Deprivation [Count of Participants; unit: Participants] — Each health authority used its own definition: Scotland used SIMD (Scottish Index of Multiple Deprivation), England used EIMD (English Index of Multiple Deprivation) and New Zealand used NZDep (New Zealand Index of Deprivation).
  Participants
    Quintile 1 (most deprived) | 455 | 393 | 848
    Quintile 2 | 484 | 511 | 995
    Quintile 3 | 505 | 499 | 1004
    Quintile 4 | 467 | 489 | 956
    Quintile 5 (least deprived) | 447 | 473 | 920
    Not recorded | 154 | 145 | 299
    Missing | 14 | 16 | 30
Clinical Management at Randomisation [Count of Participants; unit: Participants]
  CABG surgery | 81 | 80 | 161
  Drug eluting stent | 1364 | 1366 | 2730
  Bare metal stent | 13 | 14 | 27
  Medical management | 169 | 164 | 333
  Conservative | 69 | 67 | 136
  ICA planned | 830 | 835 | 1665

OUTCOME MEASURES:

1. Primary Outcome: Time-to-event: All-cause Mortality
Description: Restricted Mean Survival Time
Time Frame: Date of index MI to 15 months
Population: Intention to Treat Population. Patients were analysed according to their allocated intervention, irrespective of whether the patient's actual management complied with the allocated intervention.
Measure: Mean (Standard Error); unit: days
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
days | 447.337 (1.0542) | 445.196 (1.1741)

2. Primary Outcome: Incidence: All-cause Mortality
Description: Occurrence of event
Time Frame: Date of index MI to 15 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
Participants | 68 | 87
Statistical Analysis 1: Comparison: 3 Months Dual Anti-platelet Therapy vs 12 Months Dual Anti-platelet Therapy; The primary analysis compared the primary and secondary outcomes between groups using a Cox regression model, stratifying by country to account for clustering of participants, and adjusting for cardiac history as a fixed effect (stratification factor in randomisation). Results are reported as an adjusted hazard ratio (HR) with its corresponding 95% confidence interval (CI) and p-value; Test type: Superiority; p = 0.1232, Regression, Cox; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.57 to 1.07] — 3 versus 12 months (the comparator)

3. Secondary Outcome: Time-to-event: Non-cardiovascular Death (Including Fatal Bleeding) and Major Non-fatal Bleeding
Description: Restricted Mean Survival Time
Time Frame: Date of MI to 15 months
Population: The intention to treat (ITT) principle. Patients were analysed according to their allocated intervention, irrespective of whether the patient's actual management complied with the allocated intervention.
Measure: Mean (Standard Error); unit: days
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
days | 442.881 (1.2908) | 440.736 (1.3565)

4. Secondary Outcome: Incidence: Non-cardiovascular Death (Including Fatal Bleeding) and Major Non-fatal Bleeding
Description: Occurrence of event
Time Frame: Date of MI to 15 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
participants | 104 | 127
Statistical Analysis 1: Comparison: 12 Months Dual Anti-platelet Therapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1220, Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.63 to 1.06]

5. Secondary Outcome: Time-to-event: Non-cardiovascular Death (Including Fatal Bleeding)
Description: Restricted Mean Survival Time
Time Frame: Date of MI to 15 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
days | 452.453 (0.5873) | 452.593 (0.5285)

6. Secondary Outcome: Incidence: Non-cardiovascular Death (Including Fatal Bleeding)
Description: Occurrence of event
Time Frame: Date of MI to 15 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
participants | 27 | 29
Statistical Analysis 1: Comparison: 12 Months Dual Anti-platelet Therapy; The primary analysis compared the time to event primary and secondary outcomes between groups using a Cox regression model, stratifying by country to account for clustering of participants, and adjusting for cardiac history as a fixed effect (stratification factor in randomisation). Results are reported as an adjusted hazard ratio (HR) with its corresponding 95% confidence interval (CI) and p-value; Test type: Superiority; p = 0.7789, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.55 to 1.57]

7. Secondary Outcome: Time-to-event: Major Fatal and Non-fatal Bleeding
Description: Restricted Mean Survival Time
Time Frame: Date of MI to 15 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
days | 445.227 (1.1719) | 442.790 (1.2794)

8. Secondary Outcome: Incidence: Major Fatal and Non-fatal Bleeding
Description: Occurrence of event
Time Frame: Date of MI to 15 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
participants | 80 | 102
Statistical Analysis 1: Comparison: 12 Months Dual Anti-platelet Therapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0977, Regression, Cox; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.58 to 1.05]

9. Secondary Outcome: Time-to-event: Gastrointestinal Bleeding
Description: Restricted Mean Survival Time
Time Frame: Date of MI to 15 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
days | 449.967 (0.8887) | 450.562 (0.7774)

10. Secondary Outcome: Incidence: Gastrointestinal Bleeding
Description: Occurrence of event
Time Frame: Date of MI to 15 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
Participants | 36 | 38
Statistical Analysis 1: Comparison: 12 Months Dual Anti-platelet Therapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.8208, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.60 to 1.50]

11. Secondary Outcome: Time-to-event: Cardiovascular Death and Non-fatal Myocardial Infarction
Description: Restricted Mean Survival Time
Time Frame: Date of MI to 15 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
days | 422.876 (2.1559) | 424.670 (2.1010)

12. Secondary Outcome: Incidence: Cardiovascular Death and Non-fatal Myocardial Infarction
Description: Occurrence of event
Time Frame: Date of MI to 15 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
Participants | 236 | 226
Statistical Analysis 1: Comparison: 12 Months Dual Anti-platelet Therapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.6158, Regression, Cox; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.87 to 1.26]

13. Secondary Outcome: Time-to-event: Cardiovascular Mortality (Cardiac and Non-cardiac)
Description: Restricted Mean Survival Time
Time Frame: Date of MI to 15 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
days | 449.943 (0.8891) | 447.897 (1.0372)

14. Secondary Outcome: Incidence: Cardiovascular Mortality (Cardiac and Non-cardiac)
Description: Occurrence of event
Time Frame: Date of MI to 15 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
Participants | 40 | 56
Statistical Analysis 1: Comparison: 12 Months Dual Anti-platelet Therapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1020, Regression, Cox; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.48 to 1.07]

15. Secondary Outcome: Time-to-event: Myocardial Infarction (Fatal and Non-fatal)
Description: Restricted Mean Survival Time
Time Frame: Date of MI to 15 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
days | 424.471 (2.1157) | 427.444 (2.0181)

16. Secondary Outcome: Incidence: Myocardial Infarction (Fatal and Non-fatal)
Description: Occurrence of event
Time Frame: Date of MI to 15 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
Participants | 221 | 203
Statistical Analysis 1: Comparison: 12 Months Dual Anti-platelet Therapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3623, Regression, Cox; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.90 to 1.32]

17. Secondary Outcome: Incidence: Intracranial Haemorrhage
Description: Occurrence of event
Time Frame: Date of MI to 15 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
Participants | 0 | 10

18. Secondary Outcome: Time-to-event: Coronary Revascularisation
Description: Restricted Mean Survival Time
Time Frame: Date of MI to 15 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
days | 414.488 (2.3733) | 417.081 (2.3383)

19. Secondary Outcome: Incidence: Coronary Revascularisation
Description: Occurrence of event
Time Frame: Date of MI to 15 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
Participants | 286 | 259
Statistical Analysis 1: Comparison: 12 Months Dual Anti-platelet Therapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.2324, Regression, Cox; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.94 to 1.31]

20. Secondary Outcome: Time-to-event: Stent Thrombosis
Description: Restricted Mean Survival Time
Time Frame: Date of MI to 15 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
days | 450.566 (0.8329) | 450.026 (0.9228)

21. Secondary Outcome: Incidence: Stent Thrombosis
Description: Occurrence of event
Time Frame: Date of MI to 15 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
Participants | 34 | 32
Statistical Analysis 1: Comparison: 12 Months Dual Anti-platelet Therapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.8104, Regression, Cox; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.66 to 1.72]

22. Secondary Outcome: Time-to-event: Thrombotic Stroke
Description: Restricted Mean Survival Time
Time Frame: Date of MI to 15 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
days | 453.711 (0.4353) | 454.244 (0.3519)

23. Secondary Outcome: Incidence: Thrombotic Stroke
Description: Occurrence of event
Time Frame: Date of MI to 15 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
Participants | 13 | 7
Statistical Analysis 1: Comparison: 12 Months Dual Anti-platelet Therapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1875, Regression, Cox; Hazard Ratio (HR) = 1.86, 95% CI 2-sided [0.74 to 4.65]

24. Other Pre Specified Outcome: Time-to-event: Iron Therapy
Description: Restricted Mean Survival Time
Time Frame: Date of MI to 15 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2526 | 2526
days | 439.175 (1.5407) | 439.749 (1.4840)

25. Other Pre Specified Outcome: Incidence: Iron Therapy
Description: Occurrence of event
Time Frame: Date of MI to 15 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2265 | 2269
Participants | 116 | 122
Statistical Analysis 1: Comparison: 12 Months Dual Anti-platelet Therapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.7220, Regression, Cox; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.74 to 1.23]

26. Other Pre Specified Outcome: Time-to-event: Blood Transfusion
Description: Restricted Mean Survival Time
Time Frame: Date of MI to 15 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2164 | 2164
days | 430.118 (2.1292) | 430.346 (2.1049)

27. Other Pre Specified Outcome: Incidence: Blood Transfusion
Description: Occurrence of event
Time Frame: Date of MI to 15 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
Number analyzed (Participants) | 2164 | 2164
Participants | 138 | 140
Statistical Analysis 1: Comparison: 12 Months Dual Anti-platelet Therapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.8851, Regression, Cox; Hazard Ratio (HR) = 1.017, 95% CI 2-sided [0.804 to 1.287]

ADVERSE EVENTS:
Time Frame: 15 months from date of randomisation.
Description: As the IMPs being used in the study all have marketing authorisations AEs will not be recorded in an AE log, nor reported elsewhere. The study outcomes listed will not be recorded as SAEs and will therefore not be reported to the Sponsor. Once an Investigator becomes aware that a SUSAR has occurred in a study participant, will be reported to the sponsor immediately or within 24 hours.
Arm/Group | 3 Months Dual Anti-platelet Therapy | 12 Months Dual Anti-platelet Therapy
All-Cause Mortality (participants affected / at risk) | 68/2526 | 87/2526
Serious Adverse Events (participants affected / at risk) | 0/2526 | 0/2526
Other Adverse Events (participants affected / at risk) | 0/2526 | 0/2526

LIMITATIONS AND CAVEATS:
The major limitation is that early trial termination meant the target sample size was not achieved, leaving an underpowered trial which was unable to address its primary endpoint. The recruitment suspension due to COVID-19, and the subsequent delays in re-opening of the study sites and lack of staff capacity significantly affected recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT03252249/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT03252249/SAP_001.pdf
  • Informed Consent Form (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT03252249/ICF_002.pdf